CLINICAL TRIAL: NCT04906447
Title: Hybrid Effectiveness-Implementation Trial of Guided Relaxation and Acupuncture for Chronic Sickle Cell Disease Pain
Acronym: GRACE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Florida (Other); Duke University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ardith Doorenbos, Professor in the Department of Biobehavioral Health Science, College of Nursing, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0124; 1UG3AT011265-01 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-05-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): Participants randomized to the control arm will receive usual care
- Acupuncture (Experimental): Acupuncture treatments twice a week for five weeks
  Interventions: Other: Acupuncture
- Guided Relaxation (Experimental): Daily use of a guided relaxation app for 6 weeks
  Interventions: Behavioral: Guided Relaxation

INTERVENTIONS:
Behavioral: Guided Relaxation — Guided relaxation uses the mind to reduce pain, promote well-being, and improve physical function. Guided relaxation is a state of concentration and focused attention that gives people more control over their pain experience and its impact and an increased sense of well-being.
  Arms: Guided Relaxation
Other: Acupuncture — Acupuncture is a body-based therapy that includes the insertion of thin needles at strategic points on the body that has been proven effective for reducing pain.
  Arms: Acupuncture

SUMMARY:
The investigators will conduct a hybrid type 1 effectiveness implementation trial to assess the effectiveness of acupuncture and guided relaxation on 360 people with Sickle Cell Disease (SCD), while observing and gathering information on implementation in three health systems: University of Illinois Hospital & Health Sciences System, University of Florida Health, and Duke University Health Systems. Each serves a large population with SCD, uses EPIC as their electronic health record, and has a Clinical and Translational Science Award (CTSA), which will help speed the translation of discovery into improved patient care. During the UH3 Implementation Phase, the 3-arm, 3-site randomized controlled trial will follow a quantitative modified SMART design, a pragmatic trial that evaluates adaptive interventions where the guided relaxation and acupuncture interventions respond to patients' characteristics and evolving pain status. The investigators rely on the Consolidated Framework for Implementation Research (CFIR) to plan, execute, and evaluate associated implementation processes. The use of complementary and integrative health (CIH) therapies by those with SCD to reduce pain and opioid use, to help enable them to better cope with their pain, is well known, but there are few studies that evaluate the effectiveness of these therapies, and none that also evaluates the implementation across multiple health care systems and patient populations as this study will.

Aim 1: Determine the effectiveness of guided relaxation and acupuncture as compared to usual care in decreasing pain and opioid use for SCD patients. Hypothesis: At 6-weeks, SCD patients randomized to either CIH intervention will have a greater decrease in pain, opioid use, sleep, anxiety, depressive symptoms, and pain catastrophizing compared to SCD patients randomized to usual care.

Aim 2: Identify the best adaptive intervention for improved outcomes by documenting outcomes among adaptive intervention sequences: (1) initiate guided relaxation and switch to acupuncture for non-responders at midpoint; (2) initiate guided relaxation and continue with guided relaxation for non-responders at midpoint; (3) initiate acupuncture and switch to guided relaxation for non-responders at midpoint or (4) initiate acupuncture and continue with acupuncture for non-responders at midpoint.

Aim 3: Explore differences in response to the adaptive interventions by age and sex.

Aim 4: Identify implementation facilitators, challenges, and solutions for structures and processes that contribute to the seamless integration of CIH therapies into the 3 health systems by conducting individual interviews with participants in the intervention group who responded to the intervention and those who did not. The investigators will also conduct focus groups with hospital personnel at 4 timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease based on hemoglobin electrophoresis
* Provision of signed and dated informed consent form
* Able to speak and understand English
* Chronic pain, defined as a response of "Some days," "Most days" or "Every day" to the question, "In the past 3 months, how often have you had pain?" (Answer options: Never, Some days, Most days, Every day)
* Current pain interference using the general activity question from PEG, score ≥3 on 0-10 scale

Exclusion Criteria:

* Has had a stem cell transplant for sickle cell disease
* Current incarceration
* Any other condition that the investigator considers precludes participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pain Interference | From Baseline to 24 weeks
  Scores range from 4-20; higher scores indicate that pain is interfering with daily activities more
Pain, Enjoyment of Life and General Activity scale (PEG) | From Baseline to 24 weeks
  0-10 rating on pain intensity, enjoyment of life and general activity
PROMIS Physical Function | From Baseline to 24 weeks
  4-20 rating on the impact of pain on ability to perform normal activities; higher scores indicate greater impact of pain on physical function

SECONDARY OUTCOMES:
Generalised Anxiety Disorder Questionnaire (GAD-7) | From Baseline to 24 weeks
  Measure of Anxiety with scores ranging from 0-21. Higher scores indicate higher levels of anxiety.
Patient Health Questionnaire Depression Scale (PHQ) | From Baseline to 24 weeks
  0-24 rating of depression. 10 or greater total is considered major depression, 20 or more is severe major depression.
PROMIS sleep disturbance 8a | From Baseline to 24 weeks
  8-40 rating with higher scores indicating greater severity of sleep disturbance
Sleep duration | From Baseline to 24 weeks
  Hours a participant has slept
Pain Catastrophizing Scale (PCS) | From Baseline to 24 weeks
  0-52 scale with higher scores indicating more catastrophizing thoughts are present
Patient's Global Impression of Change (PGIC) | From Baseline to 24 weeks
  1-7 scale with higher scores indicating more improvement in pain from the patient's perspective
Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS1) | From Baseline to 24 weeks
  1-20 scale with higher score relating to more frequent substance use over the past 12 months
Gastrointestinal Constipation 9a | From Baseline to 24 weeks
  9-45 scale with higher scores indicating more severe constipation symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ardith Doorenbos, PhD, RN, FAAN, Principal Investigator — University of Illinois at Chicago
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
We will publish our results in open-source manuscripts that will be available to the public. Electronic copies of publications will be deposited in PubMed Central with proper tagging of metadata to ensure online discoverability and accessibility within four weeks of acceptance by a journal. To the extent feasible, Underlying Primary Data will be shared simultaneously with the publication and made immediately accessible through release under the Creative Commons Attribution 4.0 Generic License or an equivalent license, or otherwise dedicated to the public domain. Before submitting Underlying Primary Data, we will work with our Institutional Review Board (IRB) and Data Safety and Monitoring Board to assess the informed consent materials and to determine whether the Underlying Primary Data may be shared as contemplated in this policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared within one year of the completion of the study.
Access Criteria: The data and associated documentation will be made available to users only under a data-sharing agreement that provides for (a) a commitment to using the data only for research purposes and not to identify any individual patient; (b) a commitment to securing the data using appropriate computer technology; and (c) a commitment to destroying or returning the data after analyses are completed. Such a data-use agreement will be executed through the PIs and the University of Illinois at Chicago College of Nursing. The database can then be accessed via our secure website, in a format that can be used by a variety of statistical software packages. We will make our data and results publicly available (predominately online), so that they can easily be found.

REFERENCES:
- [Derived] Knisely MR, Rivera E, deMartelly VA, Abdulkadir A, Doorenbos AZ, Ezenwa MO, Molokie RE, Li H, Shah N, Schlaeger JM, Patil CL. Developing an Implementation Blueprint for the NIH HEAL Initiative GRACE Trial: Perspectives on Acupuncture and Guided Relaxation for Chronic Sickle Cell Disease Pain. J Integr Complement Med. 2023 Oct;29(10):683-688. doi: 10.1089/jicm.2022.0781. Epub 2023 May 15. PMID 37184905
- [Derived] Doorenbos AZ, Schlaeger JM, deMartelly VA, Burke LA, Boyd AD, Knisely MR, Leigh JW, Li H, Mandernach MW, Molokie RE, Patil CL, Steffen AD, Shah N, Ezenwa MO. Hybrid effectiveness-implementation trial of guided relaxation and acupuncture for chronic sickle cell disease pain (GRACE): A protocol. Contemp Clin Trials Commun. 2023 Jan 18;32:101076. doi: 10.1016/j.conctc.2023.101076. eCollection 2023 Apr. PMID 36852100

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04906447/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04906447/ICF_001.pdf